CLINICAL TRIAL: NCT04952688
Title: Modifications in Retinal Microvascularization With OCT- Angiography in Patients With First-line Colorectal Cancer, Treated With Targeted Anti-angiogenic Therapy.
Brief Title: Modifications in Retinal Microvascularization With Targeted Anti-angiogenic Therapy in Colorectal Cancer
Acronym: VOCANGIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A01178-31
Record Dates: First submitted 2021-06-18; First posted 2021-07-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: retina; OCT-angiography; Anti-VEGF; microvascularization; Targeted therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Inclusion
  Before Anti-VEGF treatment: opht
  Interventions: Other: OCT- Angiographie

INTERVENTIONS:
Other: OCT- Angiographie — Ophthalmological examinations

SUMMARY:
Retinal microvascularization can provide important informations to systemic vascular phenomena. The non-invasive quantitative description of the retinal vascularization is now possible by performing OCT-angiography and their image analysis software (vascular density and retinal perfusion). Systemic microvacular changes during the establishment of oncological treatment by targeted antiangiogenic therapy are little described in the literature. The objective of this pilot study is to describe the evolution of the retinal vascular density of patients with antiangiogenic drugs. In addition, the evolution of the retinal vascular density of patients on antiangiogenic drugs will study as a function of the response to the treatment and the toxicity of these treatments.

DETAILED DESCRIPTION:
The main objective of this study is to describe the change in retinal vascular density of patients with first-line colorectal cancer treated with Bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old starting first-line treatment for metastatic colorectal cancer including BEVACIZUMAB (AVASTIN®)
2. Systemic or intraocular anti-VEGF treatment naïve
3. ECOG ≤ 2

Exclusion Criteria:

1. Pregnant woman,
2. Minor patient or under legal protection
3. Person deprived of liberty or under guardianship
4. Inability to undergo medical monitoring of the trial
5. Impossibility of carrying out the OCT-A
6. Patient with a contraindication to Tropicamide 0.5% eye drops
7. Patient with a history of degenerative macular pathology, vascular macular pathology or presenting an epiretinal membrane with traction phenomenon.
8. Diabetes
9. Patient for whom it is not possible to schedule an ophthalmology consultation before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
retinal vascular density retinal vascular density | 12 month
  this measurement will be the average of the 4 quadrants (temporal, nasal, superior and inferior 24). It will be performed by PLEX Elite 9000 Swept Source OCT-A before, during and at the end of the anti-angiogenic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Audrey HENNEQUIN, Principal Investigator — Centre Georges François Leclerc
Locations (2):
- France (2):
  - Centre Georges François Leclerc, Dijon
  - CHU de Dijon, Dijon